CLINICAL TRIAL: NCT06776419
Title: the Role of cArdiac Inflammation, endoThelial Dysfunction, and FIbrosis in fabrY Disease
Acronym: RATIFY
Status: Recruiting | Type: Observational
Sponsor: Caroline Michaela Kistorp (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Caroline Michaela Kistorp, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-24052180
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Fabry Disease; Cardiovascular Diseases
Keywords: Hypertrophy; Inflammation; Myocardium; Fibrosis Myocardial; Endothelial dysfunction; Coronary Microcirculation
MeSH Terms: conditions — Fabry Disease; Cardiovascular Diseases; Hypertrophy; Myocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Fabry Disease: Patients with a genetically verified diagnosis of Fabry disease, grouped by the presence of left ventricular hypertrophy
  Interventions: Diagnostic Test: Cardiac Magnetic Ressonance Imaging; Diagnostic Test: 82Rubidium-positron emission tomography and computer-tomography
- Controls: Healthy age- and sex-matched controls
  Interventions: Diagnostic Test: Cardiac Magnetic Ressonance Imaging; Diagnostic Test: 82Rubidium-positron emission tomography and computer-tomography

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Ressonance Imaging — CMR-protocol with gadolinium contrast
  Other Names: CMR
Diagnostic Test: 82Rubidium-positron emission tomography and computer-tomography — cardiac Rb-PET protocol
  Other Names: 82Rb-PET/CT

SUMMARY:
The overall objective of this study is to investigate Fabry-related cardiomyopathy and the use of native T1-mapping, coronary microvascular function, cardiac inflammation, and cardiac injury in an effort to improve the ability to detect disease. The study aims to achieve this by:

1. Investigating the association between cardiac inflammation, fibrosis, and injury against the distribution and degree of microvascular disease in patients with Fabry disease with and without left ventricular hypertrophy (LVH) using cardiac magnetic resonance (CMR) imaging and 82Rubidium Positron emission tomography and computer tomography (82Rb-PET/CT).
2. Using an extensive, in-depth biomarker blood panel to investigate the pathological pathways associated with Fabry disease and Fabry-related cardiomyopathy.

DETAILED DESCRIPTION:
Fabry disease is a rare X-linked lysosomal disorder affecting 1:58,000 in the Danish population (males 1:85,000; females 1:44,000) [1]. A mutation in the gene encoding the enzyme alpha-gal A, an essential enzyme in normal lysosomal function, causes progressive cellular accumulation of the glycosphingolipids, especially globotriaosylceramide (Gb3). This leads to a severe disruption of cellular function. Men with a classic phenotype present with no or very low alpha-gal A-activity and develop early multi-organ involvement, especially renal and cardiac disease, resulting in a severely impaired prognosis [2]. However, both men and women can be affected in the presence of a disease-bearing mutation [2,3]. Females and men with a non-classic phenotype can also present with early organ involvement. However, their presentation is often more heterogeneous. While the classic male phenotype evidently need early initiation of therapy, the need of treatment is less clear in females and in males with a non-classic phenotype [3]. Furthermore, the incidence of new genetic variants of uncertain clinical significance, possibly indicating a Fabry diagnosis, has increased due to the general implementation of genetic screening programs [4-6]. At present, approximately 100 patients in Denmark are diagnosed with a disease-bearing mutation and followed at the Danish National Fabry Centre at Copenhagen University Hospital - Rigshospitalet. The continuing clinical challenge of who will need and when to initiate treatment necessitates close monitoring of patients at risk and, thus, a continued search for precise, reliable methods able to detect early cardiac involvement. Early initiation of therapy prior to the full manifestation of Fabry disease has shown to impede progression while evidence suggests a late initiation of treatment has reduced effects [7-10], further stressing the importance of early detection of Fabry cardiomyopathy and thus, early initiation of treatment.

Cardiomyopathy in Fabry disease In Fabry disease, the complication of greatest prognostic impact is cardiac manifestations, herein including arrhythmias, heart failure and cardiac death [2,3,11]. Although, the progressive deposition of Gb3 accounts for a maximum of 5% of total cardiac volume [12-14], a disproportionate cardiomyocyte hypertrophy, coronary wall thickening and endothelial dysfunction have been noted as general findings [12-14]. Indeed, left ventricular hypertrophy (LVH) has long been a hallmark of Fabry cardiomyopathy [15], however, the disproportionate relationship between a relatively small accumulation of Gb3 and the clinical cardiac manifestation of pronounced LVH has led to the proposal of the accumulation of Gb3 per se causes an early disruption of cellular function by pathways involving oxidative stress and inflammation [14-18]. The stress induced by Gb3 is believed to exacerbate left ventricular mass increase, cellular apoptosis, and cause the irreversible substitution of functioning tissue with reparative fibrosis. A key site and mechanism of stress and perhaps an early indicator of disease may, therefore, be found investigating changes across the vascular wall. Not only does Gb3 accumulation cause structural changes [12-14,19], Gb3 have been shown to induce the production of reactive oxygen species (ROS) through important inflammatory pathways such as transforming growth factor (TGF) β-dependent signaling, a key step in the Fabry-related vasculopathy preceding fibrosis [18]. The early structural changes in the endothelium might, therefore, tie directly to early and detrimental dysfunction [18,19].

Fabry-related cardiomyopathy and imaging As one of the most distinguishing factors of Fabry cardiomyopathy, the ability to accurately detect LVH is paramount. Recognizing the improved spatial resolution of CMR imaging, a shift from echocardiography to CMR has recently caused CMR to be recommended as part of routine clinical practice in supplement to echocardiography to improve detection of changes in left ventricular mass [15,20,21]. However, the addition of CMR-based approach has revealed several image-derived parameters of interest, which may provide insight into key aspects of the underlying mechanisms of Fabry disease, such as Gb3 accumulation, changes in fibrotic burden, and inflammation in the early stages of disease [15]. In general, Fabry cardiomyopathy often presents with low native T1 values irrespective of the presence of LVH, which have been suggested as an indirect measure of Gb3 burden [15,16,22]. In comparison, reparative fibrosis increases T1-values [15,16,22]. Furthermore, increased T2-values could be an indirect measure of inflammation [15-17], and interestingly, T2-values have been shown to decrease in concert with decreases in left ventricular mass following enzyme replacement therapy (ERT) [16,21]. Despite its promise, the overall use of T1 and T2 mapping has, however, not yet been implemented in clinical practice.

In comparison, PET/CT-based imaging has shown promise by detecting early Fabry-related changes such as coronary microvascular disease (CMD), which by itself provides important prognostic information [23]. However, use is limited due to radiation. The detection of CMD can elucidate on the progression of vascular endothelial dysfunction and may even be a key step in detecting early disease. Not only is the degree of CMD associated with the degree of LVH [24-26], of note, CMD seem to precede changes in left ventricular mass, as signs of CMD have been found irrespective of sex or the presence of LVH [24-26], suggesting its use is instrumental in detecting the early steps of Fabry-related cardiomyopathy.

Heterogeneity and regional disease progression? In Fabry, the cardiac involvement is believed to progress diffusely throughout the myocardium, with symmetric LVH as a key finding. However, of note, previous reports show great regional heterogeneity in the measured T1- and T2-values as well as regional differences using strain analysis to detect functional decline [15-17,22]. Furthermore, low T1-values, believed to be a pathognomonic feature of Fabry-associated cardiomyopathy, has been proposed to increase and pseudo-normalize with disease progression and the development of fibrosis, making the ability to account for change over time especially important [16]. CMR and PET/CT separately provide global measures of fibrosis, inflammation, and microvascular function, therefore, the combination of modalities may explain the regional differences specific to the individual patien. A combined approach may therefore provide key insights into the pathology of Fabry-associated cardiomyopathy - especially important in distinguishing early and late-stage disease.

ELIGIBILITY:
Patients with Fabry disease (1)

Inclusion Criteria:

* Male and female individuals with a genetically-verified diagnosis of Fabry disease
* ≥ 18 years of age
* Able to give informed consent

Exclusion Criteria:

* Any contraindication against a pharmacologically induced rest-stress PET/CT protocol according to local safety procedures such as acute coronary syndrome, severe bronchospasm, severe chronic obstructive pulmonary disease, cardiac arrhythmia.
* Any contraindication for MRI according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.
* Pregnancy

Age and sex-matched healthy controls (2)

Inclusion Criteria:

* ≥ 18 years of age
* Able to give informed consent

Exclusion Criteria:

* A genetically-verified diagnosis of Fabry disease.
* Family member to a patient with a genetically-verified diagnosis of Fabry disease
* Cancer expected to influence life expectancy.
* Known heart failure, previous apoplexy or previously established kidney disease.
* Initiation or change of antihypertensive therapy within 3 months of enrollment.
* Known LVH as evaluated on echocardiography
* Any contraindication for a pharmacologically induced stress PET/CT protocol according to local safety procedures such as acute coronary syndrome, severe bronchospasm, severe chronic obstructive pulmonary disease, cardiac arrhythmia.
* Any contraindication for MRI according to standard checklist used in clinical routine, including claustrophobia or metallic foreign bodies, metallic implants, internal electrical devices, or permanent makeup/tattoos that cannot be declared MR compatible.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients (adult) with genetically-verified diagnosis of Fabry disease.
  2. Age- and sex-matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in global myocardial flow reserve | 3 year change
  A between-group difference in change in global myocardial flow reserve (MFR), evaluated by 82Rb-PET/CT, comparing Fabry patients with controls irrespective of the presence of LVH.
Change in global native T1 | 3 year change
  A between-group difference in change in global native T1 evaluated by MRI, comparing Fabry patients with controls irrespective of the presence of LVH.

SECONDARY OUTCOMES:
Change in global myocardial flow reserve by group | 3 year change
  A between-group difference in change in global myocardial flow reserve (MFR) evaluated by 82Rb-PET/CT, comparing Fabry patients with controls accounting for the presence of LVH.
Change in global T1 by group | 3 year change
  A between-group difference in change in global native T1 evaluated by MRI, comparing Fabry patients with controls accounting for the presence of LVH.
Change in global T2 by group | 3 year change
  A between-group difference in change in global T2 values evaluated by MRI, comparing Fabry patients with controls accounting for the presence of LVH
Change in global T2 | 3 year change
  A between-group difference in change in global T2 values evaluated by MRI, comparing Fabry patients with controls irrespective of the presence of LVH.

OTHER OUTCOMES:
Change in regional myocardial flow reserve | 3 year change
  A between-group difference in regional MFR evaluated by 82Rb-PET/CT according to the 17-segment model
Change in regional T1 | 3 year change
  A between-group difference in regional native T1 evaluated by MRI according to the 17-segment model.
Change in regional T2 | 3 year change
  A between-group difference in regional native T2 values evaluated by MRI according to the 17-segment model.
Cross-modality association | 3 year change
  Association between regional impairment in global T1, T2 and MFR and according to the 17-segment model
Cross-modality association by reparative fibrosis | Baseline
  Association between regional impairment in T1, T2, MFR, and the placement of irreversible reparative fibrosis detected using late-gadolinium enhancement.
Cross-modality concordance in reparative fibrosis | Baseline
  Association between extent and size of irreversible reparative fibrosis detected using late-gadolinium enhancement and total perfusion defect by Rb-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Kistorp, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to national legistlative restrictions, unrestricted access to individual participant data is not possible. However, data exchange will be possible upon reasonable request under the assurance of data-management in accordance with Danish law.

REFERENCES:
- [Background] Effraimidis G, Rasmussen AK, Dunoe M, Hasholt LF, Wibrand F, Sorensen SS, Lund AM, Kober L, Bundgaard H, Yazdanfard PDW, Oturai P, Larsen VA, Fraga de Abreu VH, Enevoldsen LH, Kristensen T, Svenstrup K, Bille MB, Arif F, Mogensen M, Klokker M, Backer V, Kistorp C, Feldt-Rasmussen U. Systematic cascade screening in the Danish Fabry Disease Centre: 20 years of a national single-centre experience. PLoS One. 2022 Nov 16;17(11):e0277767. doi: 10.1371/journal.pone.0277767. eCollection 2022. PMID 36383556
- [Background] Waldek S, Patel MR, Banikazemi M, Lemay R, Lee P. Life expectancy and cause of death in males and females with Fabry disease: findings from the Fabry Registry. Genet Med. 2009 Nov;11(11):790-6. doi: 10.1097/GIM.0b013e3181bb05bb. PMID 19745746
- [Background] Wilcox WR, Oliveira JP, Hopkin RJ, Ortiz A, Banikazemi M, Feldt-Rasmussen U, Sims K, Waldek S, Pastores GM, Lee P, Eng CM, Marodi L, Stanford KE, Breunig F, Wanner C, Warnock DG, Lemay RM, Germain DP; Fabry Registry. Females with Fabry disease frequently have major organ involvement: lessons from the Fabry Registry. Mol Genet Metab. 2008 Feb;93(2):112-28. doi: 10.1016/j.ymgme.2007.09.013. Epub 2007 Nov 26. PMID 18037317
- [Background] Schiffmann R, Fuller M, Clarke LA, Aerts JM. Is it Fabry disease? Genet Med. 2016 Dec;18(12):1181-1185. doi: 10.1038/gim.2016.55. Epub 2016 May 19. PMID 27195818
- [Background] Sachdev B, Takenaka T, Teraguchi H, Tei C, Lee P, McKenna WJ, Elliott PM. Prevalence of Anderson-Fabry disease in male patients with late onset hypertrophic cardiomyopathy. Circulation. 2002 Mar 26;105(12):1407-11. doi: 10.1161/01.cir.0000012626.81324.38. PMID 11914245
- [Background] Monserrat L, Gimeno-Blanes JR, Marin F, Hermida-Prieto M, Garcia-Honrubia A, Perez I, Fernandez X, de Nicolas R, de la Morena G, Paya E, Yague J, Egido J. Prevalence of fabry disease in a cohort of 508 unrelated patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2007 Dec 18;50(25):2399-403. doi: 10.1016/j.jacc.2007.06.062. PMID 18154965
- [Background] Weidemann F, Niemann M, Stork S, Breunig F, Beer M, Sommer C, Herrmann S, Ertl G, Wanner C. Long-term outcome of enzyme-replacement therapy in advanced Fabry disease: evidence for disease progression towards serious complications. J Intern Med. 2013 Oct;274(4):331-41. doi: 10.1111/joim.12077. Epub 2013 May 6. PMID 23586858
- [Background] Weidemann F, Niemann M, Breunig F, Herrmann S, Beer M, Stork S, Voelker W, Ertl G, Wanner C, Strotmann J. Long-term effects of enzyme replacement therapy on fabry cardiomyopathy: evidence for a better outcome with early treatment. Circulation. 2009 Feb 3;119(4):524-9. doi: 10.1161/CIRCULATIONAHA.108.794529. Epub 2009 Jan 19. PMID 19153271
- [Background] Pieroni M, Camporeale A, Della Bona R, Sabini A, Cosmi D, Magnolfi A, Bolognese L. Progression of Fabry cardiomyopathy despite enzyme replacement therapy. Circulation. 2013 Oct 8;128(15):1687-8. doi: 10.1161/CIRCULATIONAHA.113.002799. No abstract available. PMID 24100483
- [Background] Rombach SM, Smid BE, Bouwman MG, Linthorst GE, Dijkgraaf MG, Hollak CE. Long term enzyme replacement therapy for Fabry disease: effectiveness on kidney, heart and brain. Orphanet J Rare Dis. 2013 Mar 25;8:47. doi: 10.1186/1750-1172-8-47. PMID 23531228
- [Background] Patel V, O'Mahony C, Hughes D, Rahman MS, Coats C, Murphy E, Lachmann R, Mehta A, Elliott PM. Clinical and genetic predictors of major cardiac events in patients with Anderson-Fabry Disease. Heart. 2015 Jun;101(12):961-6. doi: 10.1136/heartjnl-2014-306782. Epub 2015 Feb 5. PMID 25655062
- [Background] Linhart A, Elliott PM. The heart in Anderson-Fabry disease and other lysosomal storage disorders. Heart. 2007 Apr;93(4):528-35. doi: 10.1136/hrt.2005.063818. No abstract available. PMID 17401074
- [Background] Yogasundaram H, Kim D, Oudit O, Thompson RB, Weidemann F, Oudit GY. Clinical Features, Diagnosis, and Management of Patients With Anderson-Fabry Cardiomyopathy. Can J Cardiol. 2017 Jul;33(7):883-897. doi: 10.1016/j.cjca.2017.04.015. Epub 2017 May 4. PMID 28668140
- [Background] Frustaci A, Chimenti C, Doheny D, Desnick RJ. Evolution of cardiac pathology in classic Fabry disease: Progressive cardiomyocyte enlargement leads to increased cell death and fibrosis, and correlates with severity of ventricular hypertrophy‬‬‬‬‬‬‬‬. Int J Cardiol. 2017 Dec 1;248:257-262. doi: 10.1016/j.ijcard.2017.06.079. Epub 2017 Jun 23. PMID 28688718
- [Background] Esposito R, Santoro C, Mandoli GE, Cuomo V, Sorrentino R, La Mura L, Pastore MC, Bandera F, D'Ascenzi F, Malagoli A, Benfari G, D'Andrea A, Cameli M. Cardiac Imaging in Anderson-Fabry Disease: Past, Present and Future. J Clin Med. 2021 May 6;10(9):1994. doi: 10.3390/jcm10091994. PMID 34066467
- [Background] Nordin S, Kozor R, Vijapurapu R, Augusto JB, Knott KD, Captur G, Treibel TA, Ramaswami U, Tchan M, Geberhiwot T, Steeds RP, Hughes DA, Moon JC. Myocardial Storage, Inflammation, and Cardiac Phenotype in Fabry Disease After One Year of Enzyme Replacement Therapy. Circ Cardiovasc Imaging. 2019 Dec;12(12):e009430. doi: 10.1161/CIRCIMAGING.119.009430. Epub 2019 Dec 12. PMID 31826677
- [Background] Nordin S, Kozor R, Bulluck H, Castelletti S, Rosmini S, Abdel-Gadir A, Baig S, Mehta A, Hughes D, Moon JC. Cardiac Fabry Disease With Late Gadolinium Enhancement Is a Chronic Inflammatory Cardiomyopathy. J Am Coll Cardiol. 2016 Oct 11;68(15):1707-1708. doi: 10.1016/j.jacc.2016.07.741. No abstract available. PMID 27712787
- [Background] Choi JB, Seol DW, Do HS, Yang HY, Kim TM, Byun YG, Park JM, Choi J, Hong SP, Chung WS, Suh JM, Koh GY, Lee BH, Wee G, Han YM. Fasudil alleviates the vascular endothelial dysfunction and several phenotypes of Fabry disease. Mol Ther. 2023 Apr 5;31(4):1002-1016. doi: 10.1016/j.ymthe.2023.02.003. Epub 2023 Feb 8. PMID 36755495
- [Background] Pollmann S, Scharnetzki D, Manikowski D, Lenders M, Brand E. Endothelial Dysfunction in Fabry Disease Is Related to Glycocalyx Degradation. Front Immunol. 2021 Nov 30;12:789142. doi: 10.3389/fimmu.2021.789142. eCollection 2021. PMID 34917096
- [Background] Hazari H, Belenkie I, Kryski A, White JA, Oudit GY, Thompson R, Fung T, Dehar N, Khan A. Comparison of Cardiac Magnetic Resonance Imaging and Echocardiography in Assessment of Left Ventricular Hypertrophy in Fabry Disease. Can J Cardiol. 2018 Aug;34(8):1041-1047. doi: 10.1016/j.cjca.2018.03.011. Epub 2018 Mar 29. PMID 29935990
- [Background] Perry R, Shah R, Saiedi M, Patil S, Ganesan A, Linhart A, Selvanayagam JB. The Role of Cardiac Imaging in the Diagnosis and Management of Anderson-Fabry Disease. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1230-1242. doi: 10.1016/j.jcmg.2018.11.039. PMID 31272606
- [Background] Sado DM, White SK, Piechnik SK, Banypersad SM, Treibel T, Captur G, Fontana M, Maestrini V, Flett AS, Robson MD, Lachmann RH, Murphy E, Mehta A, Hughes D, Neubauer S, Elliott PM, Moon JC. Identification and assessment of Anderson-Fabry disease by cardiovascular magnetic resonance noncontrast myocardial T1 mapping. Circ Cardiovasc Imaging. 2013 May 1;6(3):392-8. doi: 10.1161/CIRCIMAGING.112.000070. Epub 2013 Apr 5. PMID 23564562
- [Background] Aljizeeri A, Ahmed AI, Suliman I, Alfaris MA, Elneama A, Al-Mallah MH. Incremental prognostic value of positron emission tomography-derived myocardial flow reserve in patients with and without diabetes mellitus. Eur Heart J Cardiovasc Imaging. 2023 Apr 24;24(5):563-571. doi: 10.1093/ehjci/jead023. PMID 36814411
- [Background] Spinelli L, Giudice CA, Riccio E, Castaldo D, Pisani A, Trimarco B. Endothelial-mediated coronary flow reserve in patients with Anderson-Fabry disease. Int J Cardiol. 2014 Dec 20;177(3):1059-60. doi: 10.1016/j.ijcard.2014.11.026. Epub 2014 Nov 5. No abstract available. PMID 25465838
- [Background] Tomberli B, Cecchi F, Sciagra R, Berti V, Lisi F, Torricelli F, Morrone A, Castelli G, Yacoub MH, Olivotto I. Coronary microvascular dysfunction is an early feature of cardiac involvement in patients with Anderson-Fabry disease. Eur J Heart Fail. 2013 Dec;15(12):1363-73. doi: 10.1093/eurjhf/hft104. Epub 2013 Jun 30. PMID 23818648
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Khawaja AZ, Cassidy DB, Al Shakarchi J, McGrogan DG, Inston NG, Jones RG. Revisiting the risks of MRI with Gadolinium based contrast agents-review of literature and guidelines. Insights Imaging. 2015 Oct;6(5):553-8. doi: 10.1007/s13244-015-0420-2. Epub 2015 Aug 8. PMID 26253982

DOCUMENTS (2):
  • Study Protocol (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT06776419/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT06776419/SAP_002.pdf